CLINICAL TRIAL: NCT03464253
Title: Transcranial Doppler Role in Prediction of Post-dural Puncture Headache in Parturients Undergoing Elective Caesarean Section
Brief Title: Prediction of Post-dural Puncture Headache in Parturients Undergoing Elective Caesarean Section
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, lecturer of Anesthesia and Surgical Intensive Care, Zagazig University
Other Study IDs: 4372/25-2-2018
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Performance of the transcranial Doppler (TCD) — Within 24 hour before the operation, TCD is performed using Siemens Acuson X300 machine with ultrasound frequency is 1 - 5 MHz probe to measure Mean Velocity and Pulsatility Index in the right middle cerebral artery.postoperatively, TCD study is performed twice at 24h and 48h after spinal anesthesia. For 5 days postoperatively, the Patients are assessed clinically for the occurrence of headache. Patients who developed PDPH will be identified and their pre and post puncture measurements will be compared with the corresponding measurements of PDPH free patients.

SUMMARY:
The parturients are at particular risk of post dural puncture headache (PDPH) because of their sex, young age, and the widespread application of spinal and epidural anesthesia. PDPH has a negative impact on quality of life, patient satisfaction, the postpartum experience with the mother's inability to bond with and care for her baby and it increases the economic burden associated with childbirth. Therefore, it is necessary to prevent or decrease its incidence and severity.

TCD enables measurement of the blood flow velocity in intracranial arteries and its parameters are affected by both fluctuations in intracranial pressure and changes in cerebral vessel diameters. The possibility of equipment mobilization, the opportunity of repeated bedside technique together with the noninvasive nature, makes TCD measurements attractive in the attempt to estimate CBF and offers potential application to predict and follow patients with PDPH.

DETAILED DESCRIPTION:
PDPH is described as severe "searing and spreading like hot metal" distributed over the occipital and frontal areas radiating to the neck and shoulders. 90% of headache will occur within three days of the procedure, and 66% within the first 48 hours. The PDPH rarely develops between 5 and 14 days after the technique however it may immediately occur after dural puncture but it is rare and should pay attention of the physician to alternative causes. The pain is increased by head movement, upright posture and relieved by lying down. It resolves either spontaneously within 7 days or within 48 h after effective treatment which is usually consists of fluid therapy, analgesics, sumatriptan and caffeine. Epidural blood patch remained the gold standard therapy but it is an invasive technique.

The exact etiology of PDPH is unknown; there is two hypothesis attempts to explain the cause. First it's known that dural tear leads to cerebrospinal fluid (CSF) leak and decreased volume of CSF result in intracranial hypotension which cause on pain sensitive intracranial structures that become stretched when assuming upright position result in pain. Second, intracranial volume is constant and equal to the sum of intracranial blood, CSF, and brain matter. After loss of CSF a compensatory reflex vasodilatation occur in the same pain sensitive blood vessels and this result in pain.

The association of common risk factors like female gender, particularly females during pregnancy, age groups of 20 - 40 years, a prior history of chronic headache, and a lower body mass index expose the patient to PDPH. The identification of factors that predict the likelihood of PDPH is important so that measures can be taken to minimize this painful complication resulting from spinal anesthesia.

Transcranial Doppler ultrasound (TCD) is a portable, safe, noninvasive and real-time tool for assessing intracranial blood hemodynamics. The first description of the technique was by Rune Aaslid in early 20th century and it has gained increasing acceptance as an accurate diagnostic and therapeutic tool in both cerebrovascular disease and neurocritical care. TCD enables measurement of the blood flow velocity in intracranial arteries and several Studies have shown that its parameters are affected by both fluctuations in intracranial pressure and changes in cerebral vessel diameters. So, as PDPH may be resulted from significant changes in cerebral blood flow, it could be visualized by TCD.

The possibility of equipment mobilization, the opportunity of repeated bedside technique together with the noninvasive nature, makes TCD measurements attractive in the attempt to estimate CBF and offers potential application to predict and follow patients with PDPH.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Pregnant female undergoing Elective caesarean section under spinal anesthesia.
* Age 18-40 years old.
* ASA I and ASA II.
* Accepted mental state of the patient.

Exclusion Criteria:

* Patient refusal.
* Contraindications to regional anesthesia as local infection, coagulopathy,….etc
* ASA Grade 3 and 4.
* Emergent caesarean section.
* Inadequate temporal window.
* Hypertensive disorders of the pregnancy.
* Atrial fibrillation.
* Significant fetal illness.
* History of allergy to local anesthetics.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant female undergoing Elective caesarean section under spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
TCD is able to predict the occurrence of PDPH in female patients undergoing spinal anesthesia for elective Caesarean Section | 5 days
  The group of patients who developed PDPH will be identified and their pre puncture cerebral blood flow measurements by TCD will be compared with the corresponding measurements of PDPH free patients to correlate the pre-puncture measurements with the occurrence of PDPH.

SECONDARY OUTCOMES:
verify that lumber puncture in PDPH patients leads to significant changes in cerebral blood flow supporting the theory of cerebral vasodilatation in PDPH patients. | 5 days
  The post-puncture TCD measurements will be compared to verify that lumber puncture and CSF leak leads to reflex vasodilatation in PDPH patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shereen E Abd Ellatif, MD, Study Director — Anesthesia and Surgical Intensive Care Department, faculty of medicine, Zagazig University; Sherif MS Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, faculty of medicine, Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD and any additional supporting information will become available starting 6 months after publication.
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Mohammed EL and El Shal SM. Efficacy of different size Quincke spinal needles in reduction of incidence of Post-Dural Puncture Headache (PDPH) in Caesarean Section (CS). Randomized controlled study. Egyptian Journal of Anaesthesia 33: 53-58, 2017
- [Background] Shah A, Bhatia PK, Tulsiani KL. Post dural puncture headache in caesarean section-a comparative study using 25G Quincke, 27G Quincke and 27G Whitacre needle. Indian J Anaesth 46(5):373-377, 2002
- [Background] Bardon J, LE Ray C, Samama CM, Bonnet MP. Risk factors of post-dural puncture headache receiving a blood patch in obstetric patients. Minerva Anestesiol. 2016 Jun;82(6):641-8. Epub 2015 Jul 29. PMID 26222393
- [Background] Sachs A, Smiley R. Post-dural puncture headache: the worst common complication in obstetric anesthesia. Semin Perinatol. 2014 Oct;38(6):386-94. doi: 10.1053/j.semperi.2014.07.007. Epub 2014 Aug 19. PMID 25146108
- [Background] Turnbull DK, Shepherd DB. Post-dural puncture headache: pathogenesis, prevention and treatment. Br J Anaesth. 2003 Nov;91(5):718-29. doi: 10.1093/bja/aeg231. PMID 14570796
- [Background] Kracoff SL and Kotlovker V. Post Dural Puncture Headache-Review and Suggested New Treatment. Open Journal of Anesthesiology 6: 148-163, 2016
- [Background] Venturelli PM, Brunser AM, Gaete J, Illanes S, Lopez J, Olavarria VV, Reccius A, Brinck P, Gonzalez F, Cavada G, Lavados PM. Reliability of Hand-Held Transcranial Doppler with M-mode Ultrasound in Middle Cerebral Artery Measurement. J Med Ultrasound. 2017 Apr-Jun;25(2):76-81. doi: 10.1016/j.jmu.2016.12.001. Epub 2017 Jan 4. PMID 30065464
- [Background] Vadhera RB, Babazade R, Suresh MS, Alvarado MC, Cruz AL, Belfort MA. Role of transcranial Doppler measurements in postpartum patients with post-dural puncture headache: a pilot study. Int J Obstet Anesth. 2017 Feb;29:90-91. doi: 10.1016/j.ijoa.2016.10.010. Epub 2016 Nov 4. No abstract available. PMID 28012860
- [Background] Nowaczewska M, Ksiazkiewicz B. Cerebral blood flow characteristics in patients with post-lumbar puncture headache. J Neurol. 2012 Apr;259(4):665-9. doi: 10.1007/s00415-011-6236-1. Epub 2011 Sep 21. PMID 21935623
- [Derived] Mowafy SMS, Abd Ellatif SE. Transcranial Doppler role in prediction of post-dural puncture headache in parturients undergoing elective cesarean section: prospective observational study. J Anesth. 2019 Jun;33(3):426-434. doi: 10.1007/s00540-019-02652-2. Epub 2019 May 9. PMID 31073654